CLINICAL TRIAL: NCT01675271
Title: Effect Of Individual Exercise Prescription On Cardiovascular Risk Factors In Woman At Risk For Gestational Diabetes - Focus On Autonomic Nervous System And Inflammation
Brief Title: Autonomic Nervous System and Exercise In Gestational Diabetes
Acronym: ANS-EXE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maritta Poyhonen-Alho, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300/E9/06
Record Dates: First submitted 2012-06-17; First posted 2012-08-29 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Gestational Diabetes; Cardiovascular Risk Factors
Keywords: gestational diabetes; inflammation; autonomic nervous system
MeSH Terms: conditions — Diabetes, Gestational; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- individual exercise (Active Comparator): individualized exercise program
  Interventions: Other: individual exercise
- general exercise (Active Comparator): general exercise program
  Interventions: Other: general exercise
- control (No Intervention): No exercise and dietary counselling

INTERVENTIONS:
Other: individual exercise — individual exercise and dietary prescription
  Arms: individual exercise
Other: general exercise — general exercise counselling
  Arms: general exercise

SUMMARY:
The focus of this study is on individualized exercise prescription on primary prevention of cardiovascular diseases (CVD). Special attention is set on autonomic nervous system function and inflammation.

This study will seek novel, cost-effective models of exercise prescription that will emphasize individuals own response on her health and which would be easily implemented to primary health care as primary prevention for CVD. According to power calculation,sixty women planning pregnancy with BMI equal or over 30 and/or history of GDM will be recruited and randomized to an individual exercise arm (n=20), a general exercise arm (n=20) and a control arm (n=20). General intervention group will receive general exercise and dietary counselling whereas a personal exercise and dietary programs will be planned for individualized exercise group. Those randomized to the control arm will receive no dietary and exercise information.

Clinical exercise tests and autonomic nervous system tests will be performed in the beginning of the study and after 3 months intervention. Blood samples for markers of inflammation, glucose homeostasis and lipid status will be collected from prepregnancy period until 1 years after delivery.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is one of the earliest signs for increased risk of developing CVD. In addition to this independent association, GDM increases CVD risk through type 2 diabetes. The physiological basis for his disease progression is not yet fully understood. Increasing evidence exists on interplay of insulin resistance and subclinical inflammation, and more recently on unbalance of the autonomic nervous system.

There is unequivocal evidence that increased physical activity and regular exercise can prevent risk factors that give rise to cardiovascular complications. According to a recent meta-analysis, exercise started before and continued throughout pregnancy may lead to marked GDM risk reduction. Unfortunately, exercise in most lifestyle studies is usually unstructured or unsupervised or does not meet current guidelines. There is also a significant gap in our understanding of how to target, deliver and prescribe the beneficial type of exercise to patients at risk in the community.

Sixty women planning pregnancy with BMI equal or over 30 and/or history of GDM will be recruited and randomized to an individual exercise arm (n=20), a general exercise arm (n=20) and a control arm (n=20). General intervention group will receive general exercise and dietary counselling whereas a personal exercise and dietary programs will be planned for individualized exercise group. Those randomized to the control arm will receive no dietary and exercise information. All subjects will be followed by diabetes nurses every 3 months as follows: at the time of recruitment, after 3 months intervention period, int the 1st, 2nd and 3rd trimester of pregnancy and 6 weeks, 6 months and 1 year postpartum. The following measurements will be performed at every visit:blood pressure, weight, waist-to-hip ratio, glucose homeostasis (2-h OGTT, Pf- insulin, Pf- glucose, insulin resistance (Homa-IR), GHbA1c, lipids (total cholesterol, LDL, HDL, triglycerides), inflammatory markers (sCRP,S-amyloid A, IL-1 and 6, alpha 1-glycoprotein, SHBG), adipokines (endothelin, adrenomedullin, adiponectin),dipeptidyl peptidase-4 (DPP-4), atrial natriuretic peptides (ANP, proBNP).For all study participants, 15 D and EDPS questionnaires are used for assessment of quality of life and mental health. Registered costs of the intervention will be calculated for cost-effectiveness analysis.

Both endurance and strength training will be included in the exercise program of the individual exercise study group. Heart rate will be monitored with heart rate belt and registered in internet-based exercise diary which can be instantly followed by the exercise professionals. This information will be used for fine-tuning of their exercise prescription during the intervention period. Diet and weight target will be planned individually by a dietician. Actualized diet will be registered in an internet-based diary instantly followed by the study dietician who will guide the subjects personally by e-mail and suggest further dietary changes if needed.

All subjects will perform an exercise test in the beginning of the study and after 3 months intervention with a step incremental protocol on a cycle ergometer until volitional fatigue. Extensive and advanced technologies will be used to monitor exercise responses, including breath-by-breath ventilation and alveolar gas exchange; exercise ECG; impedance cardiography; automatic arterial blood pressure; analysis system for heart rate variability and blood pressure variability, baroreflex sensitivity, muscle electrical activity, arterial O2 saturation and local cerebral and muscle tissue oxygenation with near-infrared spectroscopy. The autonomic nervous system measurements, including 24 hour ECG monitoring, heart rate variability assessment with controlled breathing rate, the orthostatic test and a 5 min handgrip test, will be performed during another visit to the laboratory. Total haemoglobin mass and blood volume will be determined by carbonmonoxy rebreathing method.

ELIGIBILITY:
Inclusion Criteria:

* trying to become pregnant
* BMI equal or over 30 and/or history of gestational diabetes

Exclusion Criteria:

* diagnosed diabetes
* smoking
* user of peroral glucocorticoids
* user of SSRI medication
* physical or psychological disability
* significant co-operation difficulties (e.g. insufficient language skills)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
VO2max | after 3 months training

SECONDARY OUTCOMES:
Heart rate variability | 6 weeks postpartum
autonomic nervous system function | after 3 months training
  heart rate variability, baroreflex sensitivity, handgrip test
quality of life | 1 year after delivery
  15D questionnaire
mental health | 1 year after delivery
  EDPS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aila Tiitinen, professor, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital / dept of Obstetrics and Gynecology, Helsinki, Finland

REFERENCES:
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Carr DB, Utzschneider KM, Hull RL, Tong J, Wallace TM, Kodama K, Shofer JB, Heckbert SR, Boyko EJ, Fujimoto WY, Kahn SE. Gestational diabetes mellitus increases the risk of cardiovascular disease in women with a family history of type 2 diabetes. Diabetes Care. 2006 Sep;29(9):2078-83. doi: 10.2337/dc05-2482. PMID 16936156
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Tobias DK, Zhang C, van Dam RM, Bowers K, Hu FB. Physical activity before and during pregnancy and risk of gestational diabetes mellitus: a meta-analysis. Diabetes Care. 2011 Jan;34(1):223-9. doi: 10.2337/dc10-1368. Epub 2010 Sep 27. PMID 20876206
- [Background] Poyhonen-Alho M, Viitasalo M, Nicholls MG, Lindstrom BM, Vaananen H, Kaaja R. Imbalance of the autonomic nervous system at night in women with gestational diabetes. Diabet Med. 2010 Sep;27(9):988-94. doi: 10.1111/j.1464-5491.2010.03062.x. PMID 20722671
- [Background] Poyhonen-Alho M, Ebeling P, Saarinen A, Kaaja R. Decreased variation of inflammatory markers in gestational diabetes. Diabetes Metab Res Rev. 2011 Mar;27(3):269-76. doi: 10.1002/dmrr.1170. PMID 21309051